CLINICAL TRIAL: NCT05096403
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Multicenter Study to Evaluate the Efficacy and Safety of Pegcetacoplan in Patients With Cold Agglutinin Disease (CAD)
Brief Title: A Study to Evaluate the Efficacy and Safety of Pegcetacoplan in Patients With Cold Agglutinin Disease (CAD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Sobi.PEGCET-101
Record Dates: First submitted 2021-10-15; First posted 2021-10-27 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Cold Agglutinin Disease
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune | interventions — pegcetacoplan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Pegcetacoplan Double Blind During Part A (Active Comparator): 1080 mg, subcutaneous injection, twice weekly
  Interventions: Drug: Pegcetacoplan
- Placebo Matching Pegcetacoplan-Double-blind During Part A (Placebo Comparator): Sodium acetate, subcutaneous injection, twice weekly
  Interventions: Drug: Placebo matching Pegcetacoplan
- Open-label Pegcetacoplan During Parts B and C (Active Comparator): 1080 mg, subcutaneous injection, twice weekly
  Interventions: Drug: Pegcetacoplan
- Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan During Part A) During Parts B&C (Placebo Comparator): Sodium acetate, subcutaneous injection, twice weekly
  Interventions: Drug: Placebo matching Pegcetacoplan

INTERVENTIONS:
Drug: Pegcetacoplan — Pegcetacoplan taken twice weekly as subcutaneous injection
  Other Names: Aspaveli; Empaveli
  Arms: Open-label Pegcetacoplan During Parts B and C; Pegcetacoplan Double Blind During Part A
Drug: Placebo matching Pegcetacoplan — Placebo matching pegcetacoplan taken twice weekly as subcutaneous injection
  Arms: Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan During Part A) During Parts B&C; Placebo Matching Pegcetacoplan-Double-blind During Part A

SUMMARY:
The purpose of the study is to determine the efficacy of pegcetacoplan administration compared to placebo in increasing hemoglobin (Hgb) level from baseline and avoiding transfusion in participants with primary cold agglutinin disease (CAD).

DETAILED DESCRIPTION:
This is a blind (actual treatment not disclosed to Investigator or participant) study to study pegcetacoplan in people with cold agglutinin disease. The study will consist of a 4-week screening period where selected tests will be conducted to ensure that the patient is eligible to participate in the study, followed by Part A, a 24-week blinded treatment period where the participants will receive either pegcetacoplan or a placebo treatment, looking like pegcetacoplan but with no effect. After this period, the participants will move into Part B, a 24-week period where they will all receive pegcetacoplan. Part C is a 48-week maintenance period with pegcetacoplan for all participants. After the end of treatment participants will undergo a safety follow visit about 8 weeks after last dose.

All eligible study participants will receive pegcetacoplan or placebo treatment, administered via subcutaneous infusion twice a week at home. The subcutaneous infusion requires two small needles to be inserted into the fatty layer of tissue under the skin and the investigational medication will flow into the body. Study participants and/or caregivers will be trained on home administration of pegcetacoplan.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older.
2. Diagnosis of primary CAD.
3. Hb level ≤ 9 g/dL.
4. Documented results from bone marrow biopsy within 1 year of screening
5. Either have vaccination against Streptococcus pneumoniae, Neisseria meningitidis (Types A, C, W, Y, and B), and Haemophilus influenzae (Type B) within 2 years prior to screening or agree to receive vaccination during screening.
6. Women of childbearing potential (WOCBP), defined as any women who have experienced menarche and who are NOT permanently sterile or postmenopausal, must have a negative pregnancy test at screening and agree to use protocol-defined methods of contraception for the duration of the study and 8 weeks after their last investigational medicinal product (IMP) dose.
7. Men must agree to the following for the duration of the study and 8 weeks after their last IMP dose:

   1. Avoid fathering a child.
   2. Use protocol-defined methods of contraception.
   3. Refrain from donating sperm.
8. Willing and able to give written informed consent.

Exclusion Criteria:

1. Have received other anti-complement therapies (approved or investigational) within 5 half-lives of the agent prior to randomization.
2. Treatment with rituximab monotherapy within 12 weeks prior to randomization, or rituximab combination therapies (e.g., with bendamustine, fludarabine, other cytotoxic drugs or ibrutinib) within 16 weeks prior to randomization.
3. Diagnosis of systemic lupus erythematosus or other autoimmune diseases with antinuclear antibodies.
4. History of an aggressive lymphoma or presence of a lymphoma requiring therapy.
5. Have received an organ transplant.
6. Cold agglutinin syndrome secondary to Mycoplasma pneumoniae, Epstein-Barr virus or other specific causative infection.
7. Presence or suspicion of liver dysfunction as indicated by elevated alanine aminotransferase (ALT) > 2.5 x upper limit of normal (ULN), or direct bilirubin levels > 2 x ULN.
8. Inability to cooperate with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study physician, Study Director — Swedish Orphan Biovitrum AB
Locations (44):
- United States (5):
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Lakes Research, Miami Lakes, Florida
  - University of Iowa Hospitals & Clinics - The Hemophilia Treatment Center (HTC), Iowa City, Iowa
  - Weill Cornell Medicine / NewYork Presbyterian Hospital, New York, New York
  - East Carolina University Division of Hematology/ Oncology, Greenville, North Carolina
- Medical University, Vienna, Austria
- Belgium (3):
  - Algemeen Ziekenhuis Klina, Brasschaat
  - UZ Gasthuisberg, Leuven
  - CHU de Liège, Liège
- St. Michael's Hospital, Toronto, Canada
- Helsinki University Hospital - Comprehensive Cancer Center, Helsinki, Finland
- Georgia (2):
  - "LTD Medinvest Institute of Hematology and Transfusiology ", Tbilisi
  - Ltd M. Zodelava Hematology Centre, Tbilisi
- Germany (2):
  - Universitätsklinikum Essen Klinik f. Hämatologie - Westdeutsches Tumorzentrum, Essen
  - Institut f. Transfusionsmedizin - Universität Ulm, Ulm
- Semmelweis Egyetem, Budapest, Hungary
- Italy (6):
  - A.O.R.N. S.G. Moscati di Avellino, Avellino
  - ASST degli Spedali Civili di Brescia_Presidio Ospedaliero di Brescia_U.O. Ematologia, Brescia
  - "FOND IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - AOU Maggiore della Carità SCDU Ematologia, Novara
  - Azienda Ospedaliera Ospedali Riuniti ""Villa Sofia-Cervello, Palermo
  - Grande Ospedale Metropolitano ""Bianchi - Melacrino - Morellii, Reggio Calabria
- Japan (6):
  - Fukushima Medical University Hospital, Fukushima
  - University of Tsukuba Hospital, Ibaraki
  - Ishikawa Prefectural Central Hospital, Kanazawa
  - Aichi Medical University Hospital, Nagakute
  - Shinshu University Hospital, Nagano
  - Osaka University Hospital, Osaka
- Amsterdam UMC, Amsterdam, Netherlands
- Norway (3):
  - Haukeland University Hospital, Bergen
  - Sykehuset Østfold Kalnes, Grålum
  - St Olavs Hospital, Avdeling for blodsykdommer, Trondheim
- Spain (7):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario de Gran Canaria Dr. Negrin, Las Palmas de Gran Canaria
  - Hospital Clínico Universitario de Salamanca, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico La Fe, Valencia
- United Kingdom (5):
  - St James' University Hospital, Leeds
  - Royal London Hospital, London
  - Cancer Clinical Trials Unit, Haematology -University College London -, London
  - Russell Centre for Clinical Haematology, Nottingham
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Matching Pegcetacoplan-Double-blind During Part A: Sodium acetate, subcutaneous injection, twice weekly
  Placebo matching pegcetacoplan taken twice weekly as subcutaneous injection
Period: Double-blind (Part A)
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Started | 16 | 8
Completed (Patients who completed Part A could transition into Part B.) | 14 (Patients who completed Part A could transition into Part B.) | 7 (Patients who completed Part A could transition into Part B.)
Not Completed | 2 | 1
Period: Open-label treatment (Part B)
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Started (In Part B, all patients received open-label pegcetacoplan.) | 14 (In Part B, all patients received open-label pegcetacoplan.) | 7 (In Part B, all patients received open-label pegcetacoplan.)
Completed (Patients who completed Part B could transition into Part C.) | 8 (Patients who completed Part B could transition into Part C.) | 3 (Patients who completed Part B could transition into Part C.)
Not Completed | 6 | 4
Period: Open-label maintenance period (Part C)
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Started (In Part C, all patients received open-label pegcetacoplan.) | 8 (In Part C, all patients received open-label pegcetacoplan.) | 3 (In Part C, all patients received open-label pegcetacoplan.)
Completed | 0 | 0
Not Completed | 8 | 3

BASELINE CHARACTERISTICS:
Population: All demographic characteristics are characterized by treatment group for Parts A (placebo and pegcetacoplan along with the totals) and B (total). Part A was double blinded and Part B was open-label.
Groups:
- Pegcetacoplan Double Blind During Part A: 1080 mg, subcutaneous injection, twice weekly Pegcetacoplan: Pegcetacoplan taken twice weekly as subcutaneous injection
- Placebo Matching Pegcetacoplan-Double-blind During Part A: Placebo matching pegcetacoplan taken twice weekly as subcutaneous injection
- Total: Total of all reporting groups
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A | Total
Number analyzed (Participants) | 16 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 13 | 7 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 10 | 2 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 8 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Disease History-Time since diagnosis [Mean (Standard Deviation); unit: Years] | 6.0 (5.09) | 7.0 (8.60) | 6.3 (6.30)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Achieving a Response (R) at Week 24
Description: A participant was considered to have a response if the Hgb level increased greater than or equal to (>=) 1.5 gram per deciliter (g/dL) from baseline and this increase was maintained from Week 16 through Week 24 in absence of blood transfusion from Week 5 through Week 24.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
Participants | 8 | 2

2. Secondary Outcome: Change From Baseline to Week 24 in Hemoglobin (Hgb) Level-Part A in the Absence of Intercurrent Events (ICEs).
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange) Mean change from Baseline to Week 24 in Hemoglobin (Hgb) level.
Time Frame: Week 24
Measure: Least Squares Mean (Standard Error); unit: grams per deciliter (g/dL)
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
grams per deciliter (g/dL) | 2.85 (0.306) | 1.36 (0.278)

3. Secondary Outcome: Number of Patients Achieving Transfusion Avoidance From Week 5 to Week 24-Part A
Description: Percentage of patients who did not receive a blood transfusion between Week 5 and Week 24 was assessed
Time Frame: Week 24
Population: Number of Patients Achieving Transfusion Avoidance at Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
Participants | 12 [-0.374 to 0.691] | 5 [0 to 0]

4. Secondary Outcome: Change From Baseline to Week 24 in FACT-An Scale Score (Quality of Life)-Part A in the Absence of Intercurrent Events (ICEs)
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange).
  FACT-An is used to measure quality of life (QoL) in patients with anemia. Each item is rated on a 5-point Likert scale:0=Not at all, 1=A little bit ,2=Somewhat, 3=Quite a bit, 4=Very much. Some items are reverse scored. Higher scores in this scale denote a better QoL with less impact of anemia.The total FACT-An scale score ranges from 0 to 160. The total score gives a comprehensive view of a patient's well-being. It combines the FACT-G with an Anemia subscale. FACT-G (27 items):Physical Well-Being (PWB) and Social/Family Well-Being (SWB) 14 items in total, Emotional Well-Being (EWB)-6 items,Functional Well-Being (FWB)-7 items, Anemia Subscale (AnS): 13 items. Total FACT-An score=FACT-G + Anemia Subscale=40 item
Time Frame: Week 24
Population: Part A
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
Units on a scale | 20.67 (19.175) | 16.40 (37.246)

5. Secondary Outcome: Number of Packed Red Blood Cell Transfusions Received by Patients From Week 5 to Week 24-Part A
Description: Number of blood transfusions received between Week 5 and Week 24 were assessed.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: Number of transfusions
Groups:
- Pegcetacoplan Double Blind During Part A; Placebo Matching Pegcetacoplan-Double-blind During Part A: Placebo matching pegcetacoplan taken twice weekly as subcutaneous injection
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
Number of transfusions | 1.5 (3.62) | 1.1 (2.80)

6. Secondary Outcome: Change From Baseline to Week 24 in LDH Levels-Part A in the Absence of Intercurrent Events (ICEs)
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange) Mean change from baseline to Week 24 in Lactate dehydrogenase (LDH) levels
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
U/L | -251.73 (211.312) | -82.00 (138.477)

7. Secondary Outcome: Change From Baseline to Week 24 in Haptoglobin Levels-Part A in the Absence of Intercurrent Events (ICEs)
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange).
  Mean change from baseline to Week 24 in Haptoglobin level
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
g/L | 0.31 (0.493) | 0.01 (0.020)

8. Secondary Outcome: Change From Baseline to Week 24 in Indirect Bilirubin-Part A in the Absence of Intercurrent Events (ICE)
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange).
  Mean change from baseline to Week 24 in Indirect bilirubin level
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
µmol/L | -31.55 (23.340) | 8.20 (19.325)

9. Secondary Outcome: Change From Baseline to Week 24 in ARC-Part A in the Absence of Intercurrent Events (ICEs)
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange).
  Mean change from baseline to Week 24 in Absolute reticulocyte counts (ARC).
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
10^9 cells/L | -41.17 (62.438) | -37.96 (19.891)

10. Secondary Outcome: Change From Baseline to Week 24 in D-dimer Levels-Part A in the Absence of Intercurrent Events (ICEs
Description: * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange) change from baseline to Week 24 in D-dimer levels.
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: µg/L FEU
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
µg/L FEU | -698.70 (927.480) | -1722.75 (3089.162)

11. Secondary Outcome: Normalization of Markers of Hemolysis (LDH) at Week 24-Part A
Description: Percentage of patients with LDH level within normal ranges and with an abnormal value at baseline.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 13 | 8
Participants | 5 | 1

12. Secondary Outcome: Normalization of Markers of Hemolysis (Indirect Bilirubin) at Week 24-Part A
Description: Percentage of patients with Indirect Bilirubin level within normal ranges and with an abnormal value at baseline.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 13 | 6
Participants | 9 | 1

13. Secondary Outcome: Normalization of Markers of Hemolysis (ARC) at Week 24-Part A
Description: Percentage of patients with ARC level within normal ranges and with an abnormal value at baseline.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 10 | 8
Participants | 4 | 2

14. Secondary Outcome: Normalization of Markers of Hemolysis (Haptoglobin) at Week 24-Part A
Description: Percentage of patients with haptoglobin level within normal ranges and with an abnormal value at baseline.
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 15 | 6
Participants | 4 | 0

15. Secondary Outcome: Count and Percentage of Patients With a First Normalization From Baseline by Week 24 for Haptoglobin Levels-Part A
Description: Percentage of patients with haptoglobin level normalization during the initial 24 weeks of the study
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 15 | 6
Participants | 7 | 0

16. Secondary Outcome: Count and Percentage of Patients With a First Normalization From Baseline by Week 24 for Hemoglobin Levels-Part A
Description: Percentage of patients with Hemoglobin level normalization during the initial 24 weeks of the study
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
Participants | 7 | 0

17. Secondary Outcome: Count and Percentage of Patients With a First Normalization From Baseline by Week 24 for LDH Levels-Part A
Description: Percentage of patients with LDH level normalization during the initial 24 weeks of the study
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 13 | 8
Participants | 6 | 2

18. Secondary Outcome: Count and Percentage of Patients With a First Normalization From Baseline by Week 24 for Indirect Bilirubin Levels-Part A
Description: Percentage of patients with Indirect Bilirubin level normalization during the initial 24 weeks of the study
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 13 | 6
Participants | 11 | 1

19. Secondary Outcome: Count and Percentage of Patients With a First Normalization From Baseline by Week 24 for ARC Levels-Part A
Description: Percentage of patients with ARC level normalization during the initial 24 weeks of the study
Time Frame: Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 10 | 8
Participants | 9 | 3

20. Secondary Outcome: Number of Packed Red Blood Cell Units Transfused From Week 5 to Week 24-Part A
Description: Number of PRBC units transfused from Week 5 and Week 24 was assessed
Time Frame: Week 5 to Week 24
Measure: Mean (Standard Deviation); unit: Number of PRBC units transfused
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
Number of PRBC units transfused | 2.47 (5.944) | 1.88 (4.549)

21. Secondary Outcome: Change From Baseline to Week 24 in FACIT-F Subscale Score-Part A in the Absence of Intercurrent Events (ICEs)
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange).
  The FACIT-F subscale is used to measure fatigue and its impact upon daily activities and function in patients with chronic illnesses and contains 20 items related to the impact of fatigue. Each item is scored on a 0-4 scale, with some items reverse-scored. Total scores range from 0 to 52, where higher scores indicate less fatigue and better outcomes, and lower scores reflect greater fatigue. It can be used alone or with other FACIT subscales as part of broader quality of life assessments.
Time Frame: Week 24
Population: Part A
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
Units on a scale | 9.73 (11.028) | 8.80 (18.130)

22. Secondary Outcome: Change From Baseline to Week 24 in SF-12-Part A in the Absence of Intercurrent Events (ICEs)
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange.
  SF-12 is a 12-item health survey assessing physical and mental health. Higher scores mean better health with scores above 50 indicating better than average health. It produces two summary scores: the Physical Component Summary (PCS) and Mental Component Summary (MCS), both norm-based (mean=50, SD=10), with ranges of ~5-80 (PCS) and ~-3.3-80 (MCS). Higher scores=better health. It also covers 8 subscales-Physical Functioning (PF), Role-Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role-Emotional (RE), and Mental Health (MH), each scored between 0-100, where higher=better functioning. Scores are computed using weighted formulas from item responses (not simple averages).
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
units on a scale
  Physical Component Score at Week 24 | 4.95 (7.965) | 4.46 (11.867)
  Mental Component Score at Week 24 | 5.53 (9.935) | 2.50 (9.777)

23. Secondary Outcome: Change From Baseline to Week 24 in EQ-5D-5L Questionnaire -Part A in the Absence of Intercurrent Events (ICEs)
Description: The EQ-5D-5L measures total health across 5 dimensions: Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression-each scored from 1 (no problems) to 5 (extreme problems). Scores form a 5-digit health profile (e.g., 12345). Each individual score plus a VAS for perceived health status today are separately reported. Higher scores reflect better total health. The EQ VAS is a patient-rated score from 0 (worst) to 100 (best health).
  The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange).
Time Frame: Week 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A
Number analyzed (Participants) | 16 | 8
units on a scale
  Mobility-Part A | 0.50 (1.087) | 0.00 (1.633)
  Self-care-Part A | 0.00 (0.447) | 1.00 (1.414)
  Usual activities-Part A | 0.58 (0.669) | 0.00 (0.816)
  Pain/Discomfort-Part A | 0.25 (0.866) | -0.75 (1.258)
  Anxiety/Depression-Part A | 0.33 (0.492) | 0.00 (0.816)

24. Secondary Outcome: Change From Baseline to Week 48 in Hemoglobin (Hgb) Level-Part B in the Absence of Intercurrent Events (ICEs).
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange).
  Mean change from Baseline to Week 48 in Hemoglobin (Hgb) level.
Time Frame: Week 48
Population: Part B
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Groups:
- Open-label Pegcetacoplan During Part B: 1080 mg, subcutaneous injection, twice weekly
- Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan During Part A) During Part B: Placebo matching pegcetacoplan taken twice weekly as subcutaneous injection
Arm/Group | Open-label Pegcetacoplan During Part B | Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan During Part A) During Part B
Number analyzed (Participants) | 14 | 7
grams per deciliter (g/dL) | 3.00 (2.101) | 3.35 (0.995)

25. Secondary Outcome: Change From Baseline to Week 48 in LDH Level-Part B in the Absence of Intercurrent Events (ICEs).
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange).
  Mean change from Baseline to Week 48 in LDH level.
Time Frame: Week 48
Population: Part B
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Open-label Pegcetacoplan During Part B | Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan During Part A) During Part B
Number analyzed (Participants) | 14 | 7
U/L | -220.25 (168.347) | -259.25 (52.258)

26. Secondary Outcome: Change From Baseline to Week 48 in Haptoglobin Level-Part B in the Absence of Intercurrent Events (ICEs).
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange).
  Mean change from Baseline to Week 48 in Haptoglobin level
Time Frame: Week 48
Population: Part B
Measure: Mean (Standard Deviation); unit: grams per deciliter (g/dL)
Arm/Group | Open-label Pegcetacoplan During Part B | Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan During Part A) During Part B
Number analyzed (Participants) | 14 | 7
grams per deciliter (g/dL) | 0.18 (0.238) | 0.69 (0.262)

27. Secondary Outcome: Change From Baseline to Week 48 in Indirect Bilirubin Level-Part B in the Absence of Intercurrent Events (ICEs).
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange).
  Mean change from Baseline to Week 48 in Indirect Bilirubin level.
Time Frame: Week 48
Population: Part B
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | Open-label Pegcetacoplan During Part B | Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan During Part A) During Part B
Number analyzed (Participants) | 14 | 7
µmol/L | -40.19 (28.546) | -33.43 (25.237)

28. Secondary Outcome: Change From Baseline to Week 48 in ARC-Part B in the Absence of Intercurrent Events (ICEs)
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange).
  Mean change from baseline to Week 48 in Absolute reticulocyte counts (ARC).
Time Frame: Week 48
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Open-label Pegcetacoplan During Part B | Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan During Part A) During Part B
Number analyzed (Participants) | 14 | 7
10^9 cells/L | -39.64 (55.966) | -118.20 (73.076)

29. Secondary Outcome: Change From Baseline to Week 48 in D-dimer Levels-Part B in the Absence of Intercurrent Events (ICEs).
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange).
  Mean change from baseline to Week 48 in D-dimer levels.
Time Frame: Week 48
Measure: Mean (Standard Deviation); unit: µg/L FEU
Arm/Group | Open-label Pegcetacoplan During Part B | Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan During Part A) During Part B
Number analyzed (Participants) | 14 | 7
µg/L FEU | -596.63 (937.910) | -3595.00 (4879.037)

30. Secondary Outcome: Change From Baseline to Week 48 in FACT-An Scale Score (Quality of Life)-Part B in the Absence of Intercurrent Events (ICEs)
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug and plasma exchange.
  The FACT-An is used to measure quality of life (QoL) in patients with anemia. Each item is rated on a 5-point Likert scale:0=Not at all, 1=A little bit ,2=Somewhat, 3=Quite a bit, 4=Very much.Some items are reverse scored. Higher scores in this scale denote a better QoL with less impact of anemia. The total FACT-An scale score ranges from 0 to 160. The total score gives a comprehensive view of a patient's well-being. It combines the FACT-G with an Anemia subscale.FACT-G (27 items):Physical Well-Being (PWB) and Social/Family Well-Being (SWB) 14 items in total, Emotional Well-Being (EWB)-6 items, Functional Well-Being (FWB)-7 items, Anemia Subscale (AnS): 13 items. Total FACT-An score=FACT-G + Anemia Subscale=40 items
Time Frame: Week 48
Population: Part B
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Pegcetacoplan During Part B | Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan During Part A) During Part B
Number analyzed (Participants) | 14 | 7
Units on a scale | 29.20 (19.113) | 39.50 (29.771)

31. Secondary Outcome: Change From Baseline to Week 48 in FACIT-F Subscale Score-Part B in the Absence of Intercurrent Events (ICEs).
Description: as for outcome 21
Time Frame: Week 48
Population: Part B
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Pegcetacoplan During Part B | Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan During Part A) During Part B
Number analyzed (Participants) | 14 | 7
Units on a scale | 11.82 (11.252) | 21.75 (14.315)

32. Secondary Outcome: Change From Baseline to Week 48 in EQ-5D-5L-Part B in the Absence of Intercurrent Events (ICEs).
Description: as for outcome 23
Time Frame: Week 48
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Open-label Pegcetacoplan During Part B | Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan During Part A) During Part B
Number analyzed (Participants) | 10 | 4
Units on a scale
  Mobility-Part B | 0.60 (1.174) | 1.25 (1.708)
  Self-care-Part B | 0.10 (0.316) | 1.25 (0.957)
  Usual activities-Part B | 0.70 (0.949) | 0.75 (1.258)
  Pain/Discomfort-Part B | 0.40 (0.966) | 1.00 (1.414)
  Anxiety/Depression-Part B | 0.30 (0.483) | 0.00 (1.414)

33. Secondary Outcome: Change From Baseline to Week 48 in SF-12-Part B in the Absence of Intercurrent Events (ICEs).
Description: The ICEs of interest were :
  * Withdrawal from treatment or lost to follow-up before the end of the double-blind period
  * Use of prohibited medications (rituximab alone or in combination, any other complement inhibitor, any other investigational drug, and plasma exchange SF-12 is a 12-item health survey assessing physical and mental health. Higher scores mean better health with scores above 50 indicating better than average health. It produces two summary scores: the Physical Component Summary (PCS) and Mental Component Summary (MCS), both norm-based (mean = 50, SD =10), with ranges of ~5-80 (PCS) and ~-3.3-80 (MCS). Higher scores = better health. It also covers 8 subscales-Physical Functioning (PF), Role-Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role-Emotional (RE), and Mental Health (MH), each scored between 0-100, where higher=better functioning. Scores are computed using weighted formulas from item responses (not simple averages).
Time Frame: Week 48
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Open-label Pegcetacoplan During Part B | Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan During Part A) During Part B
Number analyzed (Participants) | 10 | 4
units on a scale
  Physical Component Score at Week 48 | 7.70 (8.318) | 14.49 (9.197)
  Mental Component Score at Week 48 | 3.93 (12.465) | 4.10 (8.606)

ADVERSE EVENTS:
Time Frame: Through study completion and follow-up for up to 104 weeks (24 months approximately).
Description: All safety analyses were carried out descriptively on the safety set and presented by randomization sequence. For each output summary, all data was presented as it became available. For example, data for Part A was presented when Part A was reported. When Part B data are available, all cumulative data from Parts A and B will be reported together. The data was presented by Part A and Part B.
Groups:
- Pegcetacoplan Double Blind During Part A; Placebo Matching Pegcetacoplan-Double-blind During Part A; Open-label Pegcetacoplan During Parts B and C; Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan during Part A) During Parts B&C: Initially assigned in Part A.
Arm/Group | Pegcetacoplan Double Blind During Part A | Placebo Matching Pegcetacoplan-Double-blind During Part A | Open-label Pegcetacoplan During Parts B and C | Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan during Part A) During Parts B&C
All-Cause Mortality (participants affected / at risk) | 1/16 | 0/8 | 0/14 | 0/7
Serious Adverse Events (participants affected / at risk) | 5/16 | 1/8 | 6/14 | 1/7
Other Adverse Events (participants affected / at risk) | 16/16 | 8/8 | 12/14 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pegcetacoplan Double Blind During Part A (N=16) | Placebo Matching Pegcetacoplan-Double-blind During Part A (N=8) | Open-label Pegcetacoplan During Parts B and C (N=14) | Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan during Part A) During Parts B&C (N=7)
Covid-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Cholecystitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Syncope (General disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Breakthrough haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Cold type haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pegcetacoplan Double Blind During Part A (N=16) | Placebo Matching Pegcetacoplan-Double-blind During Part A (N=8) | Open-label Pegcetacoplan During Parts B and C (N=14) | Open-label Pegcetacoplan (Placebo Matching Pegcetacoplan during Part A) During Parts B&C (N=7)
Fatigue (General disorders) | 3 | 0 | 0 | 0
Oedema peripheral (General disorders) | 3 | 3 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 3 | 1 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 2 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Urinary Tract infection (Infections and infestations) | 0 | 1 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Cold type haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0 | 3 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Chillblains (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cold exposure injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Induration (General disorders) | 1 | 0 | 0 | 0
Injection site paraesthesia (General disorders) | 1 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 0 | 0
Injection site swelling (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Injection site mass (General disorders) | 0 | 0 | 1 | 0
Performance status decreased (General disorders) | 0 | 0 | 1 | 0
Bacteriuria (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Abdominal rigidity (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrooesophageal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Asteatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Warm autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0
Eyelid ptosis (Eye disorders) | 0 | 0 | 1 | 0
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0
Macular pseudohole (Eye disorders) | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Haemosiderosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Shoulder girdle pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Thrombin-antithrombin III complex increased (Investigations) | 1 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
Slow response to stimuli (Nervous system disorders) | 0 | 0 | 1 | 0
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cyanosis (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 0
Cardiac cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (7):
  • Study Protocol: Clinical Study Protocol v2.0 (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/03/NCT05096403/Prot_001.pdf
  • Study Protocol: Clinical Study Protocol v4.0 (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/03/NCT05096403/Prot_003.pdf
  • Study Protocol: Clinical Study Protocol v3.0 (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT05096403/Prot_002.pdf
  • Study Protocol: Clinical Study Protocol v5.0 (2023-03-13): https://cdn.clinicaltrials.gov/large-docs/03/NCT05096403/Prot_004.pdf
  • Study Protocol: Clinical Study Protocol v1.0 (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT05096403/Prot_000.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan v2.0 (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT05096403/SAP_006.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan v1.0 (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT05096403/SAP_005.pdf